CLINICAL TRIAL: NCT05431647
Title: The Effectiveness of Sensory Integration Interventions on Motor and Sensory Functions in Infants With Cortical Vision Impairment and Cerebral Palsy: A Single Blind Randomized Controlled Trial
Brief Title: Sensory Integration for Infants With Cortical Visual Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Mustafa Cemali, Phd. student, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-20/494
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Sensory Integration Disorder
Keywords: Cerebral Palsy; Cortical Visual Impairment; Sensory Integration; Motor Function; Early Intervention.
MeSH Terms: conditions — Cerebral Palsy; Blindness, Cortical

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention group: Physiotherapy and Sensory Integration Therapy (Active Comparator): Physiotherapy program
  8 weeks 2 days in a week 45 minutes per session Conventional physiotherapy
  Sensory integration therapy program
  8 weeks 2 days in a week 45 minutes per session Sensory integration therapy
  Interventions: Other: Sensory integration therapy
- Control group only Physiotherapy (Active Comparator): Physiotherapy program
  8 weeks 2 days in a week 45 minutes per session Conventional physiotherapy
  Interventions: Other: Sensory integration therapy

INTERVENTIONS:
Other: Sensory integration therapy — The individuals were divided into two as randomized controlled. Both physiotherapy and sensory integration therapy were applied to the intervention group. Each treatment was applied as 2 sessions per week, 2 days a week for 8 weeks. In the control group, only physiotherapy treatment was applied for 8 weeks, 2 days a week, 2 sessions per week.

SUMMARY:
Our study examines the effect of sensory integration training on sensory, motor and oculomotor skills in infants with cortical vision impairment .

DETAILED DESCRIPTION:
Cortical vision impairment (CVI) and Cerebral Palsy (CP) lead to decrement in sensory and motor functions of infants. The current study examined the effectiveness of sensory integration interventions on sensory, motor, and oculomotor skills in infants with cortical vision impairment. Thirty-four infants with CVI and CP aged 12-18 months were enrolled to the study. The infants were randomly divided into 2 groups as the control and intervention groups. The intervention group took sensory integration intervention 2 days a week for 8 weeks in addition to conventional physiotherapy two days a week for eight weeks. The control group only received the conventional physiotherapy program 2 days a week for 8 weeks. The duration of the treatment sessions were 45 minutes for both interventions. Before and after the intervention, sensory processing functions were evaluated with the Test of Sensory Functions in Infants (TSFI) and motor functions were evaluated with the Alberta Infant Motor Scale (AIMS).

ELIGIBILITY:
Inclusion Criteria

* Cerepral palsy
* Cortical visual impairment
* 12-18 months

Exclusion Criteria

* Not participating in treatment regularly

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-06-05 (Actual)

PRIMARY OUTCOMES:
Test of Sensory Functions in Infants (TSFI) | 30 minute
  The TSFI consists of 24 items. It was developed to evaluate sensory processing problems in infants aged 4 to 18 months. The test consists of five subsections and 24 items.
Alberta Infant Motor Scale (AIMS) | 30 minute
  The AIMS gives information about the gross motor development of infants whose corrected ages are between 0 and 18 months. In AIMS, the age of infants is calculated as the corrected age. It allows the family and the clinician to obtain information about the infant's current motor development and to compare the motor development before and after treatment.

SECONDARY OUTCOMES:
Test of Sensory Functions in Infants (TSFI) | 30 minute
  The TSFI consists of 24 items. It was developed to evaluate sensory processing problems in infants aged 4 to 18 months. The test consists of five subsections and 24 items.
Alberta Infant Motor Scale (AIMS) | 30 minute
  The AIMS gives information about the gross motor development of infants whose corrected ages are between 0 and 18 months. In AIMS, the age of infants is calculated as the corrected age. It allows the family and the clinician to obtain information about the infant's current motor development and to compare the motor development before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: mustafa cemali, Phd. student, Study Director — hacettepe üniversitesi
Locations (1):
- Occupational Therapy Department, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR